CLINICAL TRIAL: NCT00241969
Title: A Multi-Site Randomized Clinical Trial of Behavioral and Nutrition Treatment Designed to Help Preschoolers With Cystic Fibrosis Optimize Growth
Brief Title: Behavioral & Nutritional Treatment to Help CF Preschoolers Grow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DK 54915; R01DK054915 (NIH)
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis; Pancreatic Cystic Fibrosis
Keywords: nutrition therapy; preschool children; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral and Nutrition Treatment (Experimental): The behavioral and nutrition treatment combines individualized nutritional counseling that targeted increasing energy and fat intake and parent training in behavioral child-management skills based on social learning theory to improve meal-time behaviors.
  Interventions: Behavioral: Behavioral and Nutrition Treatment
- Education and Attention Control (Active Comparator): The education and attention control treatment provides education and served as a behavioral placebo in terms of controlling for attention and contact frequency provided. Families are provided with information including general nutrition, enzyme therapy, respiratory infection control, and typical child development anticipatory guidance and safety for preschool- aged children.
  Interventions: Behavioral: Education and Attention Control

INTERVENTIONS:
Behavioral: Behavioral and Nutrition Treatment — This intervention will combine individualized nutrition counseling that targets increasing energy and fat intake and parent training of effective behavioral child management skills. The treatment is delivered through 8 weekly sessions followed by 4 monthly sessions, each lasting around 60 minutes.
  Arms: Behavioral and Nutrition Treatment
Behavioral: Education and Attention Control — This intervention will provide information about a number of aspects of their child's CF care and also provides anticipatory guidance for preschoolers.The treatment is delivered through 8 weekly sessions followed by 4 monthly sessions, each lasting around 60 minutes.
  Other Names: control arm
  Arms: Education and Attention Control

SUMMARY:
The primary objective of this NIH funded clinical trial is to conduct a multi-center, randomized, controlled trial comparing two interventions: a behavioral plus nutrition intervention to a nutrition intervention. This study will (a) determine the impact of the behavioral intervention on energy intake and weight gain; (b) examine the durability of the behavioral intervention's impact on growth (weight and height) one year following treatment; and (c) explore the relation between physical activity and growth.

DETAILED DESCRIPTION:
Evidence-based nutritional interventions that achieve and sustain optimal growth in young children with cystic fibrosis (CF) do not exist, despite an urgent need. Such an intervention could positively change the course of clinical lung disease and enhance survival for these children. The primary objective of this NIH funded clinical trial is to conduct a multi-center, randomized, controlled trial comparing two interventions: a behavioral plus nutrition intervention to a nutrition (attention control) intervention. All subjects will receive nutritional care consistent with the 2001 CF Consensus Conference guidelines for pediatric nutrition.

The specific aims are to:

1. determine the impact of the behavioral intervention on energy intake and weight gain;
2. examine the durability of the behavioral intervention's impact on growth (weight and height) one year following treatment; and
3. explore the relation between physical activity and growth. The central hypothesis is that behavioral intervention will lead to better growth as measured by change in weight and height for age z scores.

From three CF Centers in Ohio, (Cincinnati Children's, Columbus Children's, Rainbow Babies and Children's Hospital in Cleveland), two referral centers in Ohio (Dayton Children's and Akron Children's), one CF Center in Michigan (University of Michigan-Ann Arbor), and one CF Center in Arizona (University of Arizona-Tucson), 100 preschoolers with CF and pancreatic insufficiency age 2 to 6 years will be randomized to one of the two conditions. The two groups will be stratified so that they are similar at the initiation of treatment on weight for age z score.

Other critical variables such as history of Pseudomonas aeruginosa infection and gender will be used as covariates in the statistical analysis plan. Outcome data (energy intake measured by 7-day diet record, weight, height) will be obtained at baseline, post-treatment (6 months), and after a 12-month follow-up (18 months post baseline).

Secondary measures will include body mass index, body composition measured by dual energy x-ray absorptiometry (DXA) and skinfolds, and growth velocity. Behavioral treatment will maximize adherence to a high energy diet and enzyme replacement therapy, and motivate children to increase their energy intake. It involves 7 weekly sessions followed by 4 monthly sessions. The attention condition controls for time of contact and number of assessments conducted.

This study advances the investigation of early nutritional interventions for young children with CF and directly addresses the need for controlled, longitudinal assessment of behavioral intervention on growth. The long-range goal is to change the standard of nutritional care for young children with CF because behavioral intervention leads to optimal growth and ultimately improves lung health and survival.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of cystic fibrosis based upon 2 of the following: a. sweat chloride by quantitative pilocarpine electrophoresis ≥60 milliequivalent/Liter (mEq/L), b. two clinical features consistent with CF, or c. genetic testing demonstrating two mutations associated with CF
* confirmation of pancreatic insufficiency based upon fecal elastase of ≤ 100 micrograms per gram of stool (or an undetectable level)
* age at enrollment to the trial of 2.0 years to 6.0 years
* at least 6 months post CF diagnosis
* consuming an unrestricted fat diet

Exclusion Criteria:

* diagnosis of developmental delay (i.e., autism, cerebral palsy, or mental retardation)
* receiving supplemental enteral nutrition via nasogastric tube, gastrostomy, or total parenteral nutrition
* diagnosed with another disease/condition (e.g., insulin dependent diabetes, congenital heart disease, significant renal disease, history of bowel resection or short bowel syndrome, colonic strictures) known to affect growth
* taking a medication (e.g., insulin, growth hormone, chronic use of systemic steroids) known to affect growth
* screening assessment shows genetic potential for height as acceptable according to the 2001 Consensus Conference guidelines and diet diary indicates daily Dietary Reference Intake (DRI) of energy average of 140% or greater (DRI of 100% will be determined as the estimated energy requirement [EER] based upon the child's age, gender, and an active physical activity level
* weight z score (age and gender adjusted) of > 1.0
* prior participation in the pilot intervention studies conducted by the PI during the prior period of R01 funding or current participation in an intervention trial conducted by the Cystic Fibrosis Therapeutics Development Network.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W. Powers, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbows and Babies Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powers SW, Piazza-Waggoner C, Jones JS, Ferguson KS, Daines C, Acton JD. Examining clinical trial results with single-subject analysis: an example involving behavioral and nutrition treatment for young children with cystic fibrosis. J Pediatr Psychol. 2006 Jul;31(6):574-81. doi: 10.1093/jpepsy/jsj049. Epub 2005 Jul 13. PMID 16014819
- [Background] Stark LJ, Opipari LC, Jelalian E, Powers SW, Janicke DM, Mulvihill MM, Hovell MF. Child behavior and parent management strategies at mealtimes in families with a school-age child with cystic fibrosis. Health Psychol. 2005 May;24(3):274-80. doi: 10.1037/0278-6133.24.3.274. PMID 15898863
- [Background] Powers SW, Patton SR, Rajan S. A comparison of food group variety between toddlers with and without cystic fibrosis. J Hum Nutr Diet. 2004 Dec;17(6):523-7. doi: 10.1111/j.1365-277X.2004.00560.x. PMID 15546429
- [Background] Mitchell MJ, Powers SW, Byars KC, Dickstein S, Stark LJ. Family functioning in young children with cystic fibrosis: observations of interactions at mealtime. J Dev Behav Pediatr. 2004 Oct;25(5):335-46. doi: 10.1097/00004703-200410000-00005. PMID 15502550
- [Background] Powers SW, Patton SR. A comparison of nutrient intake between infants and toddlers with and without cystic fibrosis. J Am Diet Assoc. 2003 Dec;103(12):1620-5. doi: 10.1016/j.jada.2003.09.024. PMID 14647088
- [Background] Powers SW, Patton SR, Byars KC, Mitchell MJ, Jelalian E, Mulvihill MM, Hovell MF, Stark LJ. Caloric intake and eating behavior in infants and toddlers with cystic fibrosis. Pediatrics. 2002 May;109(5):E75-5. doi: 10.1542/peds.109.5.e75. PMID 11986481
- [Background] Stark LJ, Jelalian E, Powers SW, Mulvihill MM, Opipari LC, Bowen A, Harwood I, Passero MA, Lapey A, Light M, Hovell MF. Parent and child mealtime behavior in families of children with cystic fibrosis. J Pediatr. 2000 Feb;136(2):195-200. doi: 10.1016/s0022-3476(00)70101-6. PMID 10657825
- [Background] Stark LJ, Mulvihill MM, Jelalian E, Bowen AM, Powers SW, Tao S, Creveling S, Passero MA, Harwood I, Light M, Lapey A, Hovell MF. Descriptive analysis of eating behavior in school-age children with cystic fibrosis and healthy control children. Pediatrics. 1997 May;99(5):665-71. PMID 9113942
- [Background] Stark LJ, Mulvihill MM, Powers SW, Jelalian E, Keating K, Creveling S, Byrnes-Collins B, Harwood I, Passero MA, Light M, Miller DL, Hovell MF. Behavioral intervention to improve calorie intake of children with cystic fibrosis: treatment versus wait list control. J Pediatr Gastroenterol Nutr. 1996 Apr;22(3):240-53. doi: 10.1097/00005176-199604000-00005. PMID 8708877
- [Background] Stark LJ, Jelalian E, Mulvihill MM, Powers SW, Bowen AM, Spieth LE, Keating K, Evans S, Creveling S, Harwood I, et al. Eating in preschool children with cystic fibrosis and healthy peers: behavioral analysis. Pediatrics. 1995 Feb;95(2):210-5. PMID 7838637
- [Background] Stark LJ, Powers SW, Jelalian E, Rape RN, Miller DL. Modifying problematic mealtime interactions of children with cystic fibrosis and their parents via behavioral parent training. J Pediatr Psychol. 1994 Dec;19(6):751-68. doi: 10.1093/jpepsy/19.6.751. PMID 7830215
- [Background] Stark LJ, Knapp LG, Bowen AM, Powers SW, Jelalian E, Evans S, Passero MA, Mulvihill MM, Hovell M. Increasing calorie consumption in children with cystic fibrosis: replication with 2-year follow-up. J Appl Behav Anal. 1993 Winter;26(4):435-50. doi: 10.1901/jaba.1993.26-435. PMID 8307828
- [Derived] Powers SW, Stark LJ, Chamberlin LA, Filigno SS, Sullivan SM, Lemanek KL, Butcher JL, Driscoll KA, Daines CL, Brody AS, Schindler T, Konstan MW, McCoy KS, Nasr SZ, Castile RG, Acton JD, Wooldridge JL, Ksenich RA, Szczesniak RD, Rausch JR, Stallings VA, Zemel BS, Clancy JP. Behavioral and nutritional treatment for preschool-aged children with cystic fibrosis: a randomized clinical trial. JAMA Pediatr. 2015 May;169(5):e150636. doi: 10.1001/jamapediatrics.2015.0636. Epub 2015 May 4. PMID 25938655
- See also: For more information on research by this team visit: — http://www.cincinnatichildrens.org/research/div/psychology/faculty-labs/powers/

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral and Nutrition Treatment: Behavioral and Nutrition Treatment
  Behavioral plus Nutrition Treatment: This intervention will combine individualized nutrition counseling that targets increasing energy and fat intake and parent training of effective behavioral child management skills.
- Education and Attention Control Treatment: Education and Attention Control Treatment
  Attention Control Treatment: This intervention will provide information about a number of aspects of their child's CF care and also provides anticipatory guidance for preschoolers.
Period: Overall Study
Arm/Group | Behavioral and Nutrition Treatment | Education and Attention Control Treatment
Started | 36 | 42
Completed | 36 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral and Nutrition Treatment | Education and Attention Control Treatment | Total
Number analyzed (Participants) | 36 | 42 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (1.2) | 3.7 (1.3) | 3.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 16 | 19 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 35 | 40 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-White | 35 | 42 | 77
Energy Intake (kcal/day) [Mean (Standard Deviation); unit: calories/day (kcal/day)] | 1462 (330) | 1461 (332) | 1462 (329)
Weight for Age Z score [Mean (Standard Deviation); unit: z-score] — Weight for age Z score was calculated using the mean measurement and the Centers for Disease Control and Prevention Anthropometric Software Program. The z score is a measure of the number of standard deviations that an observation is above or below the mean. A positive z score indicates that the observation is above the mean, a negative z score that the observation is below the mean.
  z-score | -0.36 (0.75) | -0.51 (.85) | -0.44 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Change in Energy Intake From Baseline to Post Treatment
Description: This primary outcome measure compared change in energy intake from baseline to post treatment between the behavioral and nutrition treatment and the education and attention control treatment. Energy intake was assessed using a 7-day diet diary recorded by parents and analyzed using Nutrition Data System for Research Software, Version 2011. Data were examined as average kilocalories per day over the 7 day period at baseline and post treatment. The mean (SD) change in energy intake was compared between baseline to post treatment was
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Behavioral and Nutrition Treatment | Education and Attention Control Treatment
Number analyzed (Participants) | 36 | 42
kilocalories per day | 485 (355) | 58 (248)
Statistical Analysis 1: Comparison: Behavioral and Nutrition Treatment vs Education and Attention Control Treatment; Test type: Superiority — Some data were missing for energy intake (n=3 baseline, n=13 post-treatment), thus the PROC MIXED procedure (SAS) with maximum likelihood estimation was used to analyze this outcome with time as a repeated measure factor; p < 0.001, ANCOVA; maximum likelihood estimation = 431, 95% CI 2-sided [282 to 581]; All analyses were performed on the full intention-to-treat sample (defined a priori as attending the first treatment session). Some data were missing for energy intake (N = 3 baseline; 13 post treatment), and thus the PROC MIXED procedure (SAS) with maximum likelihood estimation was used to analyze this outcome with time as a repeated measures factor, no group main effect at baseline for energy intake, and sex, baseline Pseudomonas aeruginosa status, and treatment modality as covariates in the statistical model. This model is similar to an analysis of covariance model with baseline energy intake included as an additional covariate, but the PROC MIXED model employs maximum likelihood estimation and consequently allows for data to be missing at random. The test of the time by group interaction within this PROC MIXED model indicated whether the behavioral and nutrition treatment was efficacious relative to our control treatment

2. Primary Outcome: Change in Weight for Age Z-Score (WAZ) From Baseline to Post Treatment
Description: This outcome measure examines the change in weight for age Z-score (WAZ) from baseline to post treatment. Weight was measured in kilograms, measured to the nearest 100 grams, obtained using a digital scale by trained study staff. All measurements were obtained in triplicate and then the mean used for analyses.
  Weight for age Z score was calculated using the mean measurement and the Centers for Disease Control and Prevention Anthropometric Software Program. The z score is a measure of the number of standard deviations that an observation is above or below the mean. A positive z score indicates that the observation is above the mean, a negative z score that the observation is below the mean.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Behavioral and Nutrition Treatment | Education and Attention Control Treatment
Number analyzed (Participants) | 36 | 42
z-score | 0.12 (0.40) | 0.06 (0.32)
Statistical Analysis 1: Comparison: Behavioral and Nutrition Treatment vs Education and Attention Control Treatment; Test type: Superiority — All analyses were performed on the full intention-to-treat sample (defined a priori as attending the first treatment session). Analyses of WAZ change scores were carried out within the PROC GLM procedure (SAS Institute Inc.) using an analysis of covariance model with sex, Pseudomonas aeruginosa status at baseline, treatment modality, and baseline value of the corresponding outcome variable as covariates; p = 0.25, ANCOVA; maximum likelihood = 0.09, 95% CI 2-sided [-0.06 to 0.24]; All analyses were performed on the full intention-to-treat sample (defined a priori as attending the first treatment session). Analyses of WAZ change scores were carried out within the PROC GLM procedure (SAS Institute Inc.) using an analysis of covariance model with sex, Pseudomonas aeruginosa status at baseline, treatment modality, and baseline value of the corresponding outcome variable as covariates. Group main effects on these change scores in the presence of covariates were examined to determine the efficacy of the behavioral and nutrition treatment

3. Primary Outcome: Change in Height for Age Z-Score (HAZ) From Baseline to Follow Up
Description: This outcome measure examines the change in height for age Z-score (HAZ) from baseline to follow up. Height was measured standing unless the child was unwilling to stand, then a supine measurement was obtained. All measurements were obtained in triplicate and then the mean used for analyses.
  Height for age Z score was calculated using the mean measurement and the Centers for Disease Control and Prevention Anthropometric Software Program. The z score is a measure of the number of standard deviations that an observation is above or below the mean. A positive z score indicates that the observation is above the mean, a negative z score that the observation is below the mean.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Behavioral and Nutrition Treatment | Education and Attention Control Treatment
Number analyzed (Participants) | 36 | 42
Z-score | 0.09 (0.26) | -0.02 (0.32)
Statistical Analysis 1: Comparison: Behavioral and Nutrition Treatment vs Education and Attention Control Treatment; Test type: Superiority — All analyses were performed on the full intention-to-treat sample (defined a priori as attending the first treatment session). Analyses of HAZ change scores were carried out within the PROC GLM procedure (SAS Institute Inc.) using an analysis of covariance model with sex, Pseudomonas aeruginosa status at baseline, treatment modality, and baseline value of the corresponding outcome variable as covariates; p = 0.049, ANCOVA; maximum likelihood = 0.14, 95% CI 2-sided [0.001 to 0.27]; All analyses were performed on the full intention-to-treat sample (defined a priori as attending the first treatment session). Analyses of WAZ and HAZ change scores were carried out within the PROC GLM procedure (SAS Institute Inc.) using an analysis of covariance model with sex, Pseudomonas aeruginosa status at baseline, treatment modality, and baseline value of the corresponding outcome variable as covariates. Group main effects on these change scores in the presence of covariates were examined to determine the efficacy of the behavioral and nutrition treatment

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each study visit up to the final 12 month follow up assessment (18 total months from baseline).
Arm/Group | Behavioral and Nutrition Treatment | Education and Attention Control Treatment
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/42
Other Adverse Events (participants affected / at risk) | 34/36 | 41/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Behavioral and Nutrition Treatment (N=36) | Education and Attention Control Treatment (N=42)
Digestive (Gastrointestinal disorders) | 29 | 21 — Symptoms assessed using questionnaires at each treatment session & typically reported as abdominal pain or stool issue. Clinical adjustment of enzyme replacement therapy was part of the protocol and implemented by a blinded member of the CF care team
Immune (Infections and infestations) | 12 | 19
Respiratory (Respiratory, thoracic and mediastinal disorders) | 23 | 29
Head, ears, eyes, nose, throat (Infections and infestations) | 13 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No